CLINICAL TRIAL: NCT03433170
Title: Quadrupled Semitendinosus Graft and Traditional Hamstrings Graft in Anterior Cruciate Ligament Reconstruction: Randomized Controlled Trial
Brief Title: Quadrupled Semitendinosus Graft in Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Clinica Valle del Lili (Other)
Responsible Party: Principal Investigator, Juan Pablo Martinez, Orthopaedic Surgeon, Fundacion Clinica Valle del Lili
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STX4
Record Dates: First submitted 2018-01-27; First posted 2018-02-14 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2022-10

CONDITIONS: Anterior Cruciate Ligament Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Quadrupled semitendinosus graft (Experimental): Autologous quadrupled semitendinosus graft is used to reconstruct the ACL injury
  Interventions: Procedure: Quadrupled semitendinosus graft
- ST-Gracilis graft (Active Comparator): Both gracilis and semitendinosus autologous graft are used to reconstruct the ACL injury
  Interventions: Procedure: ST-Gracilis graft

INTERVENTIONS:
Procedure: Quadrupled semitendinosus graft — Quadrupled ST graft as unique graft for the ACL reconstruction. Fixation with cortical button in femur and interference screw in tibia.
  Arms: Quadrupled semitendinosus graft
Procedure: ST-Gracilis graft — Use of both semitendinosus and gracilis graft for the ACL reconstruction. Fixation with cortical button in femur and interference screw in tibia.
  Arms: ST-Gracilis graft

SUMMARY:
Randomized controlled trial comparing reconstruction of anterior cruciate ligament (ACL) with autologous quadrupled semitendinosus graft or with both semitendinosus and gracilis. It is intended to specially evaluate if by using only the semitendinosus (ST) tendon, the strength of the limb for hamstrings is affected different compared to using both gracilis and ST.

DETAILED DESCRIPTION:
Data checks programmed by a third party after inclusion of participant number 10, 20, 30 and 42. This includes source data verification.

Simple size calculations estimating a difference of 50% in strength improvement between both groups at the six months follow-up visit. 80% power and 5% alpha error.

Strength measured with dynamometer, laxity with ACL laxity tester and function with 3 scores: IKDC, Tegner-Lysholm and KOOS.

Missing data will be minimized by double checking when registering data. It might be necessary to increase sample size to 50 patients of intermediate analysis show it is necessary to find an statistically significant difference.

Trial could be stopped early if one intervention shows to be better in the intermediate analysis. These analysis will be conducted after the first 16 and 32 participants have been included.

ELIGIBILITY:
Inclusion Criteria:

* Patients with anterior cruciate ligament injury that are candidates for surgical reconstruction with hamstrings. They should be at least 16 years old.

Exclusion Criteria:

* Multiligament injuries. Re-ruptures of the ACL.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Hamstrings Strength | 6 months
  Hamstrings strength measured with a handheld dynamometer (Lafayette model 01165 ). It is measured in Newtons.

SECONDARY OUTCOMES:
Anterior cruciate ligament rerupture | 24 months
  New ACL rupture after the surgical reconstruction. It is evaluated clinically during physical examination.
ACL laxity | 24 months
  Grade of laxity after surgery for the ACL. Measured in mm with a knee laxity measurement device (Storz).

CONTACTS AND LOCATIONS:
Overall Officials: Juan P Martinez, MD, Principal Investigator — Fundacion Clinica Valle del Lili
Locations (1):
- Fundacion Valle del Lili, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Martinez-Cano JP, Gallego A, Cuadros J, Ibarra L, Mejia FM, Velasquez-Hammerle MV, Martinez-Rondanelli A. Similar results with quadrupled semitendinosus and semitendinosus-gracilis graft in anterior cruciate ligament reconstruction: A randomised controlled trial with 2-year follow-up. J Exp Orthop. 2025 Sep 24;12(3):e70399. doi: 10.1002/jeo2.70399. eCollection 2025 Jul. PMID 41018256